CLINICAL TRIAL: NCT03142425
Title: Blood Test to Predict Radiation Response and Toxicity in Patients Undergoing Radiation Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DxTerity Diagnostics (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: DXT-RADTOX-AC02; 261201600051C-0-0-1 (NIH)
Record Dates: First submitted 2017-04-25; First posted 2017-05-05 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Radiation Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Collect blood samples and associated clinical data prior to and post radiation treatment.

DETAILED DESCRIPTION:
Exploratory study to collect paired pre- and post-irradiation blood samples from 150 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 18 or older
2. Diagnosed with a primary rectal or esophageal cancer
3. Planned radiation therapy to the esophagogastric area to a minimum of 4140 cGy for esophageal/gastroesophageal junction cancer or to pelvis to a minimum of 4500 cGy for rectal cancer as part of clinical care
4. Combining chemotherapy is allowed
5. ECOG Performance Status 0-2
6. Able to provide written informed consent

Exclusion Criteria:

1. Subjects who have received radiation within three (3) months to esophagogastric or pelvic areas prior to consent
2. Subjects, who in the opinion of the investigator, may not be able to comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients, age 18 or older, diagnosed with a primary rectal or esophageal/gastroesophageal junction cancer undergoing radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Collection of blood samples from patients prior to and post irradiation treatment. | Up to 4 months, from informed consent through follow up activities.
  Explore and validate a radiation sensitivity test for determining radiation treatment tumor response by refining and analyzing gene expression signature of blood samples collected from 150 patients prior to and post irradiation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Terbrueggen, PhD, Study Director — President and CEO
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - Kaiser Permanente Los Angeles Medical Group, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No